CLINICAL TRIAL: NCT00198185
Title: The Evaluation of Cascade PRFM on Rotator Cuff Healing
Brief Title: Cascade PRFM Study: The Evaluation of Cascade Platelet-Rich Fibrin Matrix (PRFM) on Rotator Cuff Healing
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Musculoskeletal Transplant Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 24087
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2018-01-04 (Actual); Status verified 2018-01

CONDITIONS: Rotator Cuff; Tendon Injuries
Keywords: Full Thickness Tendon Defect of Rotator Cuff
MeSH Terms: conditions — Tendon Injuries

INTERVENTIONS:
Procedure: Placement of Platelet Rich Fibrin Matrix During Arthroscopic Rotator Cuff Surgery

SUMMARY:
Hypothesis: The use of cascade platelet-rich fibrin matrix (PRFM) on medium and large sized rotator cuff tears will improve patient results versus the control results by 50%.

The purpose of this study is to examine the effect of PRFM on rotator cuff repairs. Since locally applied platelet-derived growth factor (PDGF) has shown early promise in enhancing tendon and ligament healing in anterior cruciate ligament (ACL) and medial collateral ligament (MCL) reconstruction, the investigators believe that locally applied PRFM will enhance the quality of rotator cuff repairs.

ELIGIBILITY:
Inclusion Criteria:

* Patients 45 years of age and older who have failed conservative treatment for rotator cuff pathology.
* Patients in this study will have full thickness rotator cuff tears that are classified arthroscopically as medium (1 to 3 cm) or large (3 to 5 cm) and that are treated with arthroscopic repair.

Exclusion Criteria:

* Patients who have undergone revision procedures, mini-open, or open procedures will be excluded.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-01; Primary Completion 2005-01; Study Completion 2005-01

PRIMARY OUTCOMES:
L'Insalata: preoperatively, 6 weeks, 3 months post-operatively, 12 months post-operatively
American Shoulder and Elbow Surgery (ASES) Patient Survey: preoperatively, 6 weeks, 3 months post-operatively, 12 months post-operatively

SECONDARY OUTCOMES:
Ultrasound (power Doppler imaging): 6 weeks, 3 months post-operatively
Manual muscle testing using a dynamometer: preoperatively, 3 months post-operatively, 6 months post-operatively
ASES Physician Survey: preoperatively, 3 months post-operatively, 12 months post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Russell F. Warren, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Background] Burkhart SS. Arthroscopic treatment of massive rotator cuff tears. Clin Orthop Relat Res. 2001 Sep;(390):107-18. doi: 10.1097/00003086-200109000-00013. PMID 11550856
- [Background] Burkhart SS, Danaceau SM, Pearce CE Jr. Arthroscopic rotator cuff repair: Analysis of results by tear size and by repair technique-margin convergence versus direct tendon-to-bone repair. Arthroscopy. 2001 Nov-Dec;17(9):905-12. doi: 10.1053/jars.2001.26821. PMID 11694920
- [Background] Tauro JC. Arthroscopic rotator cuff repair: analysis of technique and results at 2- and 3-year follow-up. Arthroscopy. 1998 Jan-Feb;14(1):45-51. doi: 10.1016/s0749-8063(98)70119-7. PMID 9486332
- [Background] Calvert PT, Packer NP, Stoker DJ, Bayley JI, Kessel L. Arthrography of the shoulder after operative repair of the torn rotator cuff. J Bone Joint Surg Br. 1986 Jan;68(1):147-50. doi: 10.1302/0301-620X.68B1.3941132.
- [Background] Wilson F, Hinov V, Adams G. Arthroscopic repair of full-thickness tears of the rotator cuff: 2- to 14-year follow-up. Arthroscopy. 2002 Feb;18(2):136-44. doi: 10.1053/jars.2002.30443. PMID 11830806
- [Background] Harryman DT 2nd, Mack LA, Wang KY, Jackins SE, Richardson ML, Matsen FA 3rd. Repairs of the rotator cuff. Correlation of functional results with integrity of the cuff. J Bone Joint Surg Am. 1991 Aug;73(7):982-9. PMID 1874784
- [Background] Jost B, Pfirrmann CW, Gerber C, Switzerland Z. Clinical outcome after structural failure of rotator cuff repairs. J Bone Joint Surg Am. 2000 Mar;82(3):304-14. doi: 10.2106/00004623-200003000-00002. PMID 10724223
- [Background] Gazielly DF, Gleyze P, Montagnon C. Functional and anatomical results after rotator cuff repair. Clin Orthop Relat Res. 1994 Jul;(304):43-53. PMID 8020233
- [Background] Maffulli N, Moller HD, Evans CH. Tendon healing: can it be optimised? Br J Sports Med. 2002 Oct;36(5):315-6. doi: 10.1136/bjsm.36.5.315. No abstract available. PMID 12351325
- [Background] Molloy T, Wang Y, Murrell G. The roles of growth factors in tendon and ligament healing. Sports Med. 2003;33(5):381-94. doi: 10.2165/00007256-200333050-00004. PMID 12696985
- [Background] Nakamura N, Horibe S, Matsumoto N, Tomita T, Natsuume T, Kaneda Y, Shino K, Ochi T. Transient introduction of a foreign gene into healing rat patellar ligament. J Clin Invest. 1996 Jan 1;97(1):226-31. doi: 10.1172/JCI118395. PMID 8550839
- [Background] Aspenberg P, Virchenko O. Platelet concentrate injection improves Achilles tendon repair in rats. Acta Orthop Scand. 2004 Feb;75(1):93-9. doi: 10.1080/00016470410001708190. PMID 15022816
- [Background] Weiler A, Forster C, Hunt P, Falk R, Jung T, Unterhauser FN, Bergmann V, Schmidmaier G, Haas NP. The influence of locally applied platelet-derived growth factor-BB on free tendon graft remodeling after anterior cruciate ligament reconstruction. Am J Sports Med. 2004 Jun;32(4):881-91. doi: 10.1177/0363546503261711. PMID 15150033
- [Background] Yasuda K, Tomita F, Yamazaki S, Minami A, Tohyama H. The effect of growth factors on biomechanical properties of the bone-patellar tendon-bone graft after anterior cruciate ligament reconstruction: a canine model study. Am J Sports Med. 2004 Jun;32(4):870-80. doi: 10.1177/0363546503261695. PMID 15150032
- [Background] Liu SH, Baker CL. Arthroscopically assisted rotator cuff repair: correlation of functional results with integrity of the cuff. Arthroscopy. 1994 Feb;10(1):54-60. doi: 10.1016/s0749-8063(05)80293-2. PMID 8166903
- [Background] Mafulli, N, Benazzo F. Basic Sciences of Tendons. Sports Medicine and Arthroscopy Review, 8:1-5, 2000
- [Background] Marx RE. Platelet-rich plasma (PRP): what is PRP and what is not PRP? Implant Dent. 2001;10(4):225-8. doi: 10.1097/00008505-200110000-00002. No abstract available. PMID 11813662
- [Derived] Rodeo SA, Delos D, Williams RJ, Adler RS, Pearle A, Warren RF. The effect of platelet-rich fibrin matrix on rotator cuff tendon healing: a prospective, randomized clinical study. Am J Sports Med. 2012 Jun;40(6):1234-41. doi: 10.1177/0363546512442924. Epub 2012 Apr 10. PMID 22495146